CLINICAL TRIAL: NCT00006043
Title: Phase II Trial of Temozolomide in Patients With Cisplatin-Refractory Germ Cell Tumors
Brief Title: Temozolomide in Treating Patients With Metastatic Germ Cell Tumors That Have Not Responded to Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-010; CDR0000068058 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1817
Record Dates: First submitted 2000-07-05; First posted 2004-04-02 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating patients who have metastatic germ cell tumors that have not responded to cisplatin.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of temozolomide in patients with cisplatin refractory metastatic germ cell tumors. II. Determine the safety of this treatment in these patients.

OUTLINE: Patients receive oral temozolomide on days 1-5. Treatment repeats every 28 days for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study over 25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic germ cell tumor Seminoma OR Nonseminoma Measurable disease Abnormalities on radiograph OR Alpha fetoprotein greater than 15 ng/mL OR Beta human chorionic gonadotropin greater than 2.2 mIU/L At least one measurable disease site that has not received prior radiotherapy Refractory to prior cisplatin and failed, not eligible for, or refused autologous bone marrow transplantation

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: Karnofsky 70-100% Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,000/mm3 Platelet count at lest 80,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than 1.5 times normal Transaminases no greater than 1.5 times upper limit or normal (ULN) Alkaline phosphatase no greater than 3.0 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: No medical conditions that would interfere with swallowing or cause excessive vomiting No second malignancy except basal and squamous cell skin cancer Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-02; Primary Completion 2001-11 (Actual); Study Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States